CLINICAL TRIAL: NCT05078749
Title: The Effects of Telerehabilitation Based Exercise Program in Patients With Systemic Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fulden Sarı, research assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 208
Record Dates: First submitted 2021-07-15; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis; scleroderma; telerehabilitation; exercise
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training group (Active Comparator): Continuous progressive exercise training will be applied to the treatment group. The exercises will be performed every day, twice a day, for an average of 10 minutes/session, for eight weeks. Exercise training will be updated regularly at two-week intervals. A different and progressive new exercise will be sent to the patients as a Youtube link. The patients will be interviewed by video every week.
  Interventions: Other: Exercise training group
- Control training group (Sham Comparator): The control group will be followed up as a home program by explaining the exercises and giving a brochure. They will be asked to do the exercises regularly for 7 days/week, 2 sessions/day, for eight weeks. Patients in the control group will be followed up by phone once a week.
  Interventions: Other: Control training group

INTERVENTIONS:
Other: Exercise training group — A regular advanced exercise program will be given and followed.
  Arms: Exercise training group
Other: Control training group — Basic exercises will be given at the beginning and will do the same exercises
  Arms: Control training group

SUMMARY:
Systemic Sclerosis (Ssc) is a rare, systemic autoimmune disease characterized by skin fibrosis and vasculopathy. In addition to the skin, it is a heterogeneous disease that affects multiple organs, including the musculoskeletal, cardiac, pulmonary, and gastrointestinal systems. Patients may experience many symptoms such as pain, fatigue, dyspnea, impaired hand function, dry mouth, and difficulty sleeping. As a result of these symptoms, these patients may experience a decrease in activities of daily living, physical activity level and quality of life, while psychological problems such as anxiety and depression may increase. In addition to medical treatment, rehabilitation programs for the patient are an important part of treatment to eliminate or reduce these symptoms and their consequences.

Many problems such as time and resource constraints, transportation problems prevent access and compliance with the rehabilitation program. Also; For the coronavirus disease 2019 (COVID-19) epidemic that emerged in Wuhan, China in 2019, many countries have implemented many practices such as social distance, mandatory quarantine and transportation restrictions in order to better control the spread of the virus. Many people with SSc are at risk of serious complications from COVID-19 if infected due to lung involvement (>40% have interstitial lung disease) and widespread use of immunosuppressant drugs. Most countries have recommended that people with medical conditions such as SSc undergo strict isolation during the COVID-19 pandemic. As a result, patients' access to the rehabilitation program became more difficult in this process. In addition, social isolation due to the COVID-19 outbreak may increase physical inactivity and cause complications that may develop accordingly.

When the literature was examined, no studies were found showing the effect of telerehabilitation program on anxiety depression, physical activity, sleep, fatigue and quality of life in patients with SSc.

DETAILED DESCRIPTION:
According to sample size calculation 26 patients scheduled for systemic sclerosis will be included. Patients planned for systemic sclerosis will be evaluated twice at the beginning and at the end of the 8th week. The study was planned as a prospective randomized controlled study. Patients will be randomized using a computer program and divided into two groups as telerehabilitation treatment and home exercise group. For the telerehabilitation group, a progressive exercise program video link will be sent over the internet every 2 weeks. The exercise brochure will be explained and sent to the patient group followed up with the home program only at the beginning of the program.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65
* Being literate
* Patients who received standard medical treatment and whose general condition has been stable for the last 6 months
* Having minimum smartphone or computer usage knowledge or having an acquaintance who knows this information and can help with this
* Having a computer and active internet connection at home
* Disease duration between 1 and 10 years
* Agree to participate in the study

Exclusion Criteria:

* Patients who cannot cooperate with the assessment
* Those who have orthopedic problems or neurological diseases that prevent them from doing the exercises
* Those who received treatment in a physiotherapy and rehabilitation program before
* Patients with another inflammatory disease
* Female patients who are pregnant
* Patients who have had COVID-19
* Those with a diagnosis of pulmonary arterial hypertension (PAH)
* Exercise is contraindicated for those with heart disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Evaluation Scale-Pain | First day
  The Numeric Rating Scale (NRS) was used to determine the pain level of the patients at rest, activity and at night. Patients are asked to mark the numbers between 0 and 10 at the time of assessment, in terms of rest, activity and night pain. 10 score describe severe pain while 0 score is no pain
Modified Medical Research Council Dyspnea Scale | First day
  Assessment of dyspnea was assessed with the Modified Medical Research Council (MMRC) dyspnea scale. The MMRC is a category scale consisting of 5 statements about dyspnea, scored between 0-4. As the score obtained by the patient increases, the complaint of dyspnea increases.
Multidimensional Assessment of Fatigue Scale | First day
  Fatigue assessment will be evaluated with the Turkish Version of the Multidimensional Fatigue Scale (MAF-T). The MAF-T is a 4-dimensional questionnaire that assesses the degree and severity of fatigue, the amount, duration, and type of distress it causes. According to their answers, the patients score at least 1 (no fatigue) and 50 (severe fatigue) points from the test.
International Physical Activity Questionnaire-short form | First day
  Physical activity level was evaluated with Turkish valid and reliable International Physical Activity (IPAQ) questionnaire. The questionnaire consisting of 7 questions gives information about the time spent in walking, moderate-to-vigorous and vigorous activities. The time spent sitting is considered as a separate question. A score is obtained in total score metabolic equivalent (MET)-minutes. According to the result, physical activity level is classified as 'inactive', 'minimally active' and 'very active'.
Pittsburgh sleep quality index | First day
  Sleep will be assessed by the Pittsburgh sleep quality index (PUKI). The questionnaire consists of a total of 24 questions; The first 19 questions are answered by the person, and the last 5 questions are answered by the person's family or roommate. The total score of the questionnaire varies between 0-21. The higher the PUKI score, the worse the sleep quality is. A total PUKI score of < 5 indicates 'good' sleep quality, and a total PUKI score of ≥ 5 indicates 'poor' sleep quality.
Hospital Anxiety and Depression Scale | First day
  A valid and reliable Turkish Hospital Anxiety and Depression Scale (HADS) was used to determine the anxiety and depression levels of the patients. In the questionnaire consisting of a total of 14 questions, odd-numbered questions assess anxiety and even-numbered questions assess depression. It has two subgroups, anxiety (HADS-A) and depression (HADS-D). The lowest score that patients can get from both subgroups is 0, and the highest score is 21.
Nottingham Health Profile | First day
  Quality of life will be assessed with the Turkish version of the Notthingham Health Profile (NSP) scale. NSP evaluates the physical, social and emotional health problems perceived by the patient at that moment in 2 parts. Each subgroup is scored between 0-100 in itself. The total score of the NSP questionnaire is between 0-600. A high score indicates poor quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Deran OSKAY, Prof, Study Director — Gazi University
Locations (1):
- Gazi University, Çankaya, Ankara, Turkey (Türkiye)